CLINICAL TRIAL: NCT06418724
Title: Neoadjuvant PD-1 Inhibitor and EGFR Inhibitor in Locally Advanced Cutaneous Squamous Cell Carcinoma
Acronym: NEOPECS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02.23
Record Dates: First submitted 2024-04-12; First posted 2024-05-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Cutaneous Squamous Cell Carcinoma
Keywords: immunotherapy; neoadjuvant therapy; PD-1 inhibitor; EGFR inhibitor; cetuximab; cemiplimab
MeSH Terms: interventions — Cetuximab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cetuximab and Cemiplimab (Experimental): All patients will be administered the same treatment combination.
  Cemiplimab will be administered 350mg intravenously every 21 days. A maximum of 4 cycles will be given.
  Cetuximab will be administered 400mg/m2 loading dose on day 1 and 250mg/m2 on day 8 and day 15 for a 21 day cycle for first cycle. Cetuximab will be administered 250mg/m2 on day 1, 8 and 15 for a 21 day cycle for subsequent cycles for 4 cycles.
  Interventions: Drug: Cetuximab; Drug: Cemiplimab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab is a monoclonal antibody against epidermal growth factor receptor (EGFR). EGFR is over-expressed in many human cancers, including colorectal cancers.
  Other Names: Erbitux
Drug: Cemiplimab — Cemiplimab is a fully human immunoglobulin G4 (IgG4) monoclonal antibody that binds to the programmed cell death-1 (PD-1) receptor and blocks its interaction with its ligands programmed death-ligand 1 (PD-L1) and programmed death-ligand 2 (PD-L2). Engagement of PD-1 with its ligands PD-L1 and PD-L2, which are expressed by antigen presenting cells and may be expressed by tumour cells and/or other cells in the tumour microenvironment, results in inhibition of T cell function such as proliferation, cytokine secretion, and cytotoxic activity. Cemiplimab potentiates T cell responses, including antitumour responses, through blockade of PD-1 binding to PD-L1 and PD-L2 ligands.
  Other Names: Libtayo

SUMMARY:
The NEOPECS trial is a phase II prospective, single-arm, non-randomised interventional trial for patients with borderline resectable locally advanced cutaneous squamous cell carcinoma with a 6-participant safety lead in to ensure safety of the combination in the neoadjuvant setting across 3 sites in Australia.

DETAILED DESCRIPTION:
As cutaneous squamous cell carcinoma typically occurs on sun-exposed areas of the head and neck, surgical resection of advanced disease can have significant morbidity and disfigurement and strategies to downstage disease prior to surgery, improve chance of R0 resection and reduce the risk of post-surgical relapse remain an area of need.

This study aims to determine the preliminary activity and tolerability of neo-adjuvant combination cemiplimab and cetuximab in unresectable locally advanced cutaneous squamous cell carcinoma by clinical downstaging rate to resectable status.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age and able to comply with treatment, assessment and follow up
2. Documentation of a locally advanced cutaneous squamous cell carcinoma diagnosis as evidenced by histopathology with available archival tissue. Locally Advanced cutaneous Squamous Cell Carcinoma (LASCC) defined as borderline resectable for surgery due to multiple recurrences, prior radiotherapy, large extension, bone erosion and/or deep infiltration beyond the subcutaneous tissue into muscle/nerve or, where curative resection may lead to unacceptable complications, morbidity or deformity, and ineligible for curative radiotherapy
3. Measurable disease in accordance with iRECIST criteria OR clinically measurable disease >1cm by caliper measurement. Patients with synchronous primary cutaneous squamous cell carcinoma (cSCC) tumours will be eligible.
4. Adequate bone marrow function with haemoglobin >100g/L, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L). Blood transfusion is allowable.
5. Adequate hepatic function with total bilirubin levels <1.5 upper limit normal range and Alanine aminotransferase (ALT) and AST levels <2.5 level normal range.
6. Adequate renal function with eGFR estimated with Cockcroft Gault formula >50mL/min. Serum potassium levels 3.5 - 5.5 mmoL/L, Serum magnesium levels 0.7 - 1.05 mmol/L, Serum corrected calcium levels 2.15 - 2.55 mmol/L
7. Adequate performance status of Eastern Cooperative Oncology Group (ECOG) 0-1 as assessed by investigator
8. Life expectancy of >6 months
9. Able to provide written informed consent obtained from patient and ability for patient to comply with the requirements of the trial.

Exclusion Criteria:

1. Distant metastatic disease (M1) including visceral or distant nodal metastases
2. Prior receipt of checkpoint inhibitor therapy or anti-EGFR therapy for LASCC or any other malignancy
3. Uncontrolled medical/psychiatric co-morbidity as per investigator that may jeopardize the ability of the patient to undergo trial procedures with reasonable safety
4. Uncontrolled autoimmune disease requiring active immune-suppression within 1 year of enrolment
5. Corticosteroid use of >10mg daily of oral prednisone within 2 weeks of Cycle 1 Day 1 (C1D1)
6. Known history of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases.
7. Uncontrolled infection with human immunodeficiency virus, hepatitis B, or hepatitis C infection; or has a diagnosis of immunodeficiency
8. Transplant recipient
9. Hepatitis C virus (HCV) and hepatitis B virus (HBV) testing will be performed at screening
10. Controlled HIV infection (undetectable viral load (HIV RNA PCR) and Cluster of differentiation 4 (CD4) counts above 350 either spontaneously or on a stable antiviral regimen) is permitted. Monitoring will be performed per local standards.
11. Controlled hepatitis B antibody positive infection (HBsAg+) is permitted providing a serum hepatitis B virus DNA PCR that is below the limit of detection and patient is receiving anti-viral therapy for hepatitis B. Periodic monitoring of HBV DNA is required. Anti-viral therapy for at least 6 months post the last dose of investigational study drug is required.
12. Controlled hepatitis C virus antibody positive (HCV Ab+) is permitted (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy).
13. History of another malignancy within 5 years prior to trial registration. A past history of adequately treated carcinoma-in-situ, basal cell carcinoma of skin, or superficial transitional cell carcinoma of the bladder is permitted. Patients with a history of other malignancies are eligible if they have been continuously disease free for at least 3 years after definitive primary treatment and low expected risk of recurrence.
14. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with trial protocol and follow-up schedule, including alcohol and drug abuse.
15. Pregnancy, lactation or inadequate contraception. Women must be post-menopausal, infertile or willing to use reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must have been surgically sterilized or willing to use double barrier contraception.
16. Sexually active men and women of childbearing potential who are unwilling to practice highly effective contraception prior to the start of the first treatment, during the study, and for at least 6 months after the last dose of investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Preliminary activity | 3 months
  The primary preliminary activity endpoint will be the achievement of clinical downstaging from borderline resectable status to either resectable status or surgery avoidance due to complete metabolic response with no residual pathological disease as deemed by Multi-Disciplinary Team (MDT) consensus evaluation following up to 4 cycles of neoadjuvant therapy.

SECONDARY OUTCOMES:
Treatment safety and feasibility as assessed by NCI CTCAE v5 | 12 months
  Safety and feasibility by assessment of Common Terminology Criteria for Adverse Events (CTCAE) V5.0 with the incidence of ≥ Grade 3 adverse events, < Grade 3 adverse events and SAEs and AEs leading to study treatment discontinuation.
Treatment safety and feasibility as assessed by rate of R0 resection | 12 months
  Safety and feasibility by assessment of change in rate of R0 resection. R0 resection is defined no residual tumour in surgically removed specimen of curative intent per local and central pathology review.
Pathological response rate | 12 months
  Preliminary efficacy by assessment of pathological response rate, including complete (0% residual tumour cells) and major (0-10% residual tumour cells) pathological responses, by blinded central pathology review. Complete pathological response (pCR) defined as absence of viable tumor cells in surgical specimen. Major pathological response (MPR) defined as 0-10% viable tumor cells in surgical specimen.
Overall response rate (ORR) | 12 months
  Preliminary efficacy by assessment of overall response rate (ORR) as per Modifed Response Evaluation Criteria in Solid Tumors for immune based therapeutics (iRECIST) criteria or investigator caliper assessment where disease is un-measurable by CT or MRI modalities
Progression free survival (PFS) | 12 months
  Preliminary efficacy by assessment of 12-month and median PFS using the Kaplan-Meier method. PFS is defined as the interval from date of registration to the date of first evidence of disease progression or death, whichever occurs first.
Event-free survival (EFS) | 12 months
  Preliminary efficacy by assessment of 12-month and median EFS using the Kaplan-Meier method. EFS is defined as the interval from date of registration to progressive disease or adverse events precluding surgery, inability to undergo complete (R0) resection, disease recurrence or death from any cause.
Overall survival (OS) | 12 months
  Preliminary efficacy by assessment of 12-month and median OS using the Kaplan-Meier method. OS is defined as the interval from date of registration to date of death from any cause, or the date of last known follow-up alive.
Change in predicted difficulty of surgical resection and repair | 3 months
  Change in predicted difficulty of surgical resection and repair pre- and post-neoadjuvant therapy as measured with paired surgeon-rated scaling "scale for predicted operability of cutaneous SCC". Scale scores range from Inoperable disease (A) to Complete response (F)

OTHER OUTCOMES:
To explore the relationship between cancer-immune cell-stroma interactions using spatial transcriptomics and single cell RNA sequencing and outcome. | 3 months
  To explore the relationship between cancer-immune cell-stroma interactions using spatial transcriptomics and single cell RNA sequencing and outcome.
Patient reported outcomes as assessed by EORTC QLQ-C30 | 36 months
  The European Organization for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30) will be utilized to assess the quality of life of cancer patients measured from 0-4 (Not at all - Very Much).
Patient reported outcomes as assessed by FoP-Q-SF | 36 months
  The Fear-of-Progression Questionnaire - Short Form (FoP-Q-SF) will be utilized to assess fear of cancer progression measured from 1-5 (never - very often).

CONTACTS AND LOCATIONS:
Overall Officials: Jia (Jenny) Liu, MD, PhD, FRACP, Study Chair — Kinghorn Cancer Centre/St Vincent's Hospital